CLINICAL TRIAL: NCT05489185
Title: "Randomized, Double-blind Clinical Trial to Assess the Efficacy of Tranexamic Acid in Reducing Blood Loss in Patients With Hip Fracture"
Brief Title: Clinical Trial to Assess the Efficacy of Tranexamic Acid in Reducing Blood Loss in Hip Fracture Patients.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Biogipuzkoa Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2020_TRANEXAMICO
Record Dates: First submitted 2022-08-01; First posted 2022-08-05 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2022-08

CONDITIONS: Hip Fractures
Keywords: Hip Fracture; Blood loss; tranexamic acid
MeSH Terms: conditions — Hip Fractures; Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Extracapsular fracture with intravenous contraindication (control). (Placebo Comparator): Physiological saline
  Interventions: Other: Physiologic saline
- Extracapsular fracture with intravenous contraindication (experimental). (Experimental): Amchafibrin
  Interventions: Drug: Tranexamic acid
- Extracapsular fracture without intravenous contraindication (control). (Placebo Comparator): Physiological saline
  Interventions: Other: Physiologic saline
- Extracapsular fracture without intravenous contraindication (experimental). (Experimental): Amchafibrin
  Interventions: Drug: Tranexamic acid
- Intracapsular fracture with intravenous contraindication (control). (Placebo Comparator): Physiological saline
  Interventions: Other: Physiologic saline
- Intracapsular fracture with intravenous contraindication (experimental). (Experimental): Amchafibrin
  Interventions: Drug: Tranexamic acid
- Intracapsular fracture without intravenous contraindication (control). (Active Comparator): Physiological saline
  Interventions: Other: Physiologic saline
- Intracapsular fracture without intravenous contraindication (experimental). (Experimental): Amchafibrin
  Interventions: Drug: Tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid — Intravenous or topical administration
  Arms: Extracapsular fracture with intravenous contraindication (experimental).; Extracapsular fracture without intravenous contraindication (experimental).; Intracapsular fracture with intravenous contraindication (experimental).; Intracapsular fracture without intravenous contraindication (experimental).
Other: Physiologic saline — Placebo
  Arms: Extracapsular fracture with intravenous contraindication (control).; Extracapsular fracture without intravenous contraindication (control).; Intracapsular fracture with intravenous contraindication (control).; Intracapsular fracture without intravenous contraindication (control).

SUMMARY:
Hip fracture in elderly patients is a pathology with a high economic and health impact on the patient himself and on the National Health System, especially considering the significant aging of the population of the Basque Country. Despite advances, hip fracture remains in the clinical groups with the highest in-hospital mortality. Hip fracture is associated with numerous adverse events and high mortality.

Numerous antifibrinolytics, such as tranexamic acid (TXA), have been used to limit bleeding in orthopedic surgery and thus prevent the need for blood transfusion. Numerous studies have shown that the use of tranexamic acid does not increase the risk of thrombosis.

It is proposed to carry out clinical research with drugs without commercial interest. A randomized, double-blind clinical trial to assess the efficacy of tranexamic acid in reducing blood loss in elderly patients with hip fracture.

DETAILED DESCRIPTION:
Prevention and treatment of bleeding due to general or local fibrinolysis

ELIGIBILITY:
Inclusion Criteria:

* Patients over or equal to 65 years of age, of both sexes, who are going to be operated on for a hip fracture
* Accept participation in the study (informed consent that will be signed by the patient or family member/legal representative depending on the patient's degree of autonomy).

Exclusion Criteria:

* Under treatment with another experimental drug (who is not participating in another clinical trial with an experimental drug).
* The refusal of the patient or their relatives/legal representative to participate in the study.
* Known allergy to TXA ( Hipersensivity to TXA o to any of the excipients).
* Patients with a history of seizures.
* Patients with severe renal and hepatic insufficiency.
* Patients with venous thrombosis.
* Patients with active concomitant bleeding of renal origin.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 644 (Estimated)
Dates: Start 2023-05-30 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Blood transfusion | From date of randomization until the date of hospital discharge, it is estimated to be day 3 post - operation.
  Transfusion rate from patient admission to hospital discharge.

SECONDARY OUTCOMES:
Total blood loss | From date of randomization until the date of hospital discharge, it is estimated to be day 3 post - operation.
Adverse events | 3,6,9 and 12 months
Days at hospital | From date of randomization until the date of hospital discharge, it is estimated to be day 3 post - operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Asociación Instituto Biodonostia, San Sebastián, Guipuzcoa, Spain